CLINICAL TRIAL: NCT03320616
Title: A Phase 1, Open-Label, Randomized, 4-Way Crossover Study in Subjects With Chronic Hepatitis B Virus Infection to Assess Pharmacokinetics (Fasted/Fed), Safety, Tolerability and Pharmacodynamics of Single Oral Doses of Farnesoid X Receptor Agonist EYP001a
Brief Title: EYP001a Food Effect Study in Subjects With Chronic Hepatitis B Virus (HBV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-102; 2016-004713-27 (EudraCT Number)
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: The subjects will be randomized to 1 of 4 treatment sequences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): 4 single doses of EYP001a: Period 1 first dose morning fasted, second dose morning fed; Period 2 first dose evening fasted, second dose evening fed
  Interventions: Drug: EYP001a
- Sequence 2 (Experimental): 4 single doses of EYP001a: Period 1 first dose evening fasted, second dose evening fed; Period 2 first dose morning fasted, second dose morning fed
  Interventions: Drug: EYP001a
- Sequence 3 (Experimental): 4 single doses of EYP001a: Period 1 first dose morning fed, second dose morning fasted; Period 2 first dose evening fed, second dose evening fasted
  Interventions: Drug: EYP001a
- Sequence 4 (Experimental): 4 single doses of EYP001a: Period 1 first dose evening fed, second dose evening fasted; Period 2 first dose morning fed, second dose morning fasted
  Interventions: Drug: EYP001a

INTERVENTIONS:
Drug: EYP001a — Oral EYP001a capsules - 100 mg strength

SUMMARY:
The farnesoid X receptor (FXR) regulates hepatitis B virus replication through the bile acids pathway. EYP001a is a selective, synthetic FXR agonist under development for the treatment of hepatitis B.

This Phase 1 study is designed primarily to assess Pharmacokinetics (PK) under fed and fasted conditions, and to assess the safety, tolerability and Pharmacodynamics (PD) of single oral doses of EYP001a in subjects with chronic HBV infection.

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, 4-way crossover study.

A total of 14 chronic HBV subjects will participate. Subjects will receive 4 single dose administrations of EYP001a during the study. There will be 2 separate dosing periods: 1 period with 2 single administrations of EYP001a in the morning, once under fasted conditions and once under fed condition (separated by 48.5 hours), and 1 period with 2 single administrations of EYP001a in the evening, once under fasted conditions and once under fed condition (separated by 48.5 hours).

The subjects will be randomized to 1 of 4 treatment sequences:

* Sequence 1: Period 1 first dose morning fasted, second dose morning fed; Period 2 first dose evening fasted, second dose evening fed.
* Sequence 2: Period 1 first dose evening fasted, second dose evening fed; Period 2 first dose morning fasted, second dose morning fed.
* Sequence 3: Period 1 first dose morning fed, second dose morning fasted; Period 2 first dose evening fed, second dose evening fasted.
* Sequence 4: Period 1 first dose evening fed, second dose evening fasted; Period 2 first dose morning fed, second dose morning fasted.

Participation will include an eligibility screening period of maximally 40 days, clinic stay during the treatment periods, and a followup visit 4 to 6 days after the last study drug administration.

The safety and tolerability of EYP001a will be assessed by evaluating vital signs, ECGs, liver ultrasound, clinical laboratory and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Has given voluntary written informed consent before performance of any study related procedure
2. Has documented chronic HBV infection (documented within 12 months of screening visit), with criteria at screening: hepatitis B surface antigen (HBsAg) ≥ 50 IU/mL; HBV DNA > 100 IU/mL; hepatitis Be antigen (HBeAg) negative or positive
3. Gender: male or female
4. Age: 18-65 years, inclusive, at screening
5. Body mass index (BMI): 17.0-35.0 kg/m2 inclusive, at screening
6. Weight: >60 kg for males and >45 kg for females
7. Has clinical chemistry, hematology, coagulation and urinalysis tests within normal, allowable limits (with the exception of alanine aminotransferase (ALAT) [see inclusion criterion #10]); if there is an out of range value, it must be considered clinically insignificant in order to be eligible
8. Has normal vital signs after at least 5 minutes resting in supine position at screening: 95 mm Hg < systolic blood pressure < 140 mm Hg; 45 mm Hg < diastolic blood pressure < 90 mm Hg; 40 bpm < heart rate < 90 bpm
9. Has no clinically significant abnormal 12-lead automatic electrocardiogram (ECG) (incomplete right bundle branch block can be accepted) at screening: 120 ms < PR-interval < 210 ms, QRS-duration < 120 ms, corrected QT interval (QTc) (Fridericia's) ≤ 450 msec for males and females
10. Has ALAT ≤ 3 x upper limit of normal (ULN) at screening
11. Has documented liver histology with Metavir score (F0, F1, F2 or F3) or liver fibrosis documented with non-invasive alternatives to liver biopsy (Fibroscan) or shear wave elastography (Aixplorer) value < 14.6 kPa
12. Agrees to abstain from all medication, including non-prescription and prescription medication (including vitamins and natural or herbal remedies, e.g. St. John's Wort) for 28 days prior to (each) admission to the clinical research center until discharge, except for authorized medications such as hormonal contraceptives for females (registered in The Netherlands) and paracetamol. On a case-by-case basis, regular co-medication either as defined on the separate medication exception list or as documented by written approval from the Sponsor and the PI as acceptable prior to randomization, will not be considered as a deviation from this criterion. All other situations related to co-medications are considered as deviations
13. At screening, females must be non-pregnant and non-lactating, or of non-childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year postmenopausal [amenorrhoea duration of 12 consecutive months); non-pregnancy will be confirmed for all females by a serum pregnancy test conducted at screening and at (each) admission to the clinical research center
14. Female subjects of child-bearing potential, with a fertile male sexual partner, should be willing to use adequate contraception from screening until 90 days after the followup visit. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject, is acceptable
15. Male subjects, if not surgically sterilized, should be willing to use adequate contraception and not donate sperm from (first) admission to the clinical research center until 90 days after the follow-up visit. Adequate contraception for the male subject (and his female partner) is defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the subject is acceptable
16. At screening, has no recent (<3 months) history of any clinically significant conditions, which, in the opinion of the PI, would jeopardize the safety of the subject or impact the validity of the study results
17. Willingness to abstain from alcohol and methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) from 48 hours prior to (each) admission to the clinical research center

Exclusion Criteria:

1. Previous participation in the current study
2. Employee of PRA or the Sponsor
3. Currently receives or has received during the 60 days (or 5 half-lives of the specific drug, whichever is longer) before (first) admission to the clinical research center until (the last) discharge a nucleos(t)ide-analogue therapy or other anti HBV treatment (interferons, experimental anti HBV drugs or vaccines)
4. Coinfection with hepatitis C virus (HCV), hepatitis D virus (HDV) or human immunodeficiency virus (HIV)
5. Receives or plans to receive systemic immunosuppressive medications during the study or ≤2 months prior to the first study drug administration
6. Receiving or planning to receive interferon (IFN) during the study or ≤12 months prior to the first study drug administration
7. Has significant immunosuppression from, but not limited to immunodeficiency conditions such as common variable hypogammaglobulinemia
8. Clinical diagnosis of substance abuse with alcohol (regular alcohol consumption >21 units [men] and >14 units [women] per week [1 unit = ½ pint of beer, 25 mL shot of 40% spirit or a 125 mL glass of wine]), narcotics, or cocaine ≤12 months prior to screening
9. Has any known pre-existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings.
10. Has a history of clinically significant gastrointestinal disease, especially peptic ulcerations, gastrointestinal bleeding, ulcerative colitis, cholecystectomy, Crohn's disease or Irritable Bowel Syndrome, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, or cardiovascular disease or any other condition which, in the opinion of the PI, would jeopardize the safety of the subject or impact the validity of the study results
11. Has had acute diarrhea or constipation in the 7 days before (first) admission to the clinical research center. Diarrhea will be defined as the passage of liquid feces and/or a stool frequency of > 3 times per day. Constipation will be defined as a failure to open the bowels more frequently than every other day.
12. Has a history of long QT syndrome
13. Has participated in a drug study within 30 days prior to the first drug administration in the current study
14. Has a positive drug and alcohol screen (opiates, methadone, cocaine, methamphetamines, amphetamines, ecstasy, barbiturates, benzodiazepines, tricyclic antidepressants, phencyclidine and alcohol)
15. Any current or previous (ie, ≤12 months prior to screening) abuse of drugs such as opiates, cocaine, ecstasy, or intravenous amphetamines. Subjects who admit to occasional use of cannabis will not be excluded as long as they are able to abstain from cannabis when they are in the clinical research center.
16. Has an uncontrolled current illness (e.g., active infection)
17. Has had major surgery within 30 days prior to the first drug administration, or 12 months prior to the first drug administration for gastrointestinal surgery
18. Has lost more than 100 mL of blood within 60 days prior to the first drug administration
19. Has a history of relevant drug and/or food allergies
20. Smokes more than 20 cigarettes per day
21. Non-willingness to consume the Food and Drug Administration (FDA) breakfast
22. Poor venous accessibility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Type and frequencies of adverse events | Day 1 of Period 1 through Day 7 to Day 9 of Period 2

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of EYP001a | Predose to 48 hours after dosing
  ng/mL
Time to attain maximum observed plasma concentration (Tmax) after EYP001a administration | Predose to 48 hours after dosing
  h
Area under the plasma concentration-time curve (AUC) | Predose to 48 hours after dosing
  ng*h/mL
Bile acid precursor C4 (7α hydroxy-4-cholesten-3-one) | Predose to 48 hours after dosing
  ng/mL
Bile-regulating fibroblast growth factor 19 (FGF-19) | Predose to 48 hours after dosing
  pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen van de Wetering, MD, Principal Investigator — PRA-EDS
Locations (1):
- PRA-EDS, Groningen, Netherlands